CLINICAL TRIAL: NCT00430040
Title: Vascular Benefits of Adding CarvedilolCR to Type2 Diabetic Patients on ACEI:Effects on Oxidative Stress and Inflammation.
Brief Title: Vascular Benefits of Adding CarvedilolCR to Type2 Diabetic Patients on ACEI.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1918
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: Type 2 Diabetes Mellitus; Hypertension; Carvedilol CR; Beta-blocker; Oxidative stress; Inflammation; Vascular benefits
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Inflammation | interventions — Carvedilol; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- carvedilol (Experimental): carvedilol
  Interventions: Drug: Carvedilol Controlled Release (CR); Drug: lisinopril
- lisinopril (Active Comparator): lisinopril
  Interventions: Drug: lisinopril

INTERVENTIONS:
Drug: Carvedilol Controlled Release (CR) — lisinopril starting dose in all patients 10 mg QD for 1 week then increase to 20 mg QD throughout the study.
  Initial dose: Carvedilol CR (20 mg QD, dose level 1) Titration: If tolerated, increase the dosage to 20 mg QD, 40 mg QD, and 80mg QD orally over successive intervals of at least 2 weeks to achieve target blood pressure sSBP <130 and sDBP < 80
  Other Names: COREG CR
  Arms: carvedilol
Drug: lisinopril — lisinopril starting dose in all patients 10 mg QD for 1 week then increase to 20 mg QD throughout the study
  Other Names: lisinopril 10mg

SUMMARY:
To determine whether addition of Carvedilol CR to diabetic patients with hypertension who are receiving the ACEi,Lisinopril,will provide added benefits to blood vessels when compared to treatment with Lisinopril alone.It is believed that carvedilol provides added benefits by suppressing free radicals(charged substances that cause damage to the body ) and inflammation.

DETAILED DESCRIPTION:
Type 2 diabetes is an atherosclerotic, pro-inflammatory and pro-oxidative stress.Both vascular oxidative stress and inflammation are CVD risk factors and impact endothelial function.

Carvedilol has been demonstrated in preclinical and clinical studies (although limited in size) to exert anti-inflammatory and antioxidant properties: (1) reduce the inflammation markers such as high sensitivity C-reactive protein (hsCRP); (2) reduce oxidative stress via dually eliminating existing reactive oxygen species (ROS) and suppressing the generation of ROS; (3) prevent lipid peroxidation in myocardial cell membrane; (4) protect endothelial and vascular muscle cells from oxygen radical-mediated injury.

This project is about studying the effect of carvedilol CR on blood vessels of diabetic hypertensive patients as compared to Lisinopril alone.

This study involves weaning patient off their current antihypertensive medications and starting them on Lisinopril with Carvedilol CR or lisinopril alone for 6 months and studying the effects of the drugs during this period and thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female >= 18 and <= 70 years of age
* Has a documented history of type 2 diabetes mellitus for a minimum of four months prior to the screening visit
* Has a documented history of or current presentation with Stage 1 or Stage 2 hypertension and meets one of the following criteria:
* Has controlled hypertension (sSBP <130 mmHg AND sDBP <80 mmHg) on >=2 antihypertensive medications NOTE: A combination drug containing two antihypertensive agents represents two antihypertensive medications OR
* Has uncontrolled hypertension (sSBP >=130 and <=170 mmHg AND/OR sDBP >=80 and <=105 mmHg) on one or two antihypertensive medications OR
* Has newly diagnosed or previously untreated hypertension (sSBP >=130 and <=170 mmHg AND/OR sDBP >=80 and <=105 mmHg
* At Randomization, sitting systolic blood pressure (sSBP) >= 130 mmHg or sitting diastolic blood pressure (sDBP) >= 80 mmHg and sSBP <= 170 mmHg and sDBP <= 105 mmHg
* Has been on a stable dose of a 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitor (statin) for a minimum of four months prior to the screening visit

Exclusion Criteria:

* Has any clinically significant abnormality identified in the screening physical examination, laboratory tests or electrocardiogram which, in the judgement of the investigator, would preclude safe completion of the study
* Is female of childbearing potential
* Has any of these cardiac conditions: uncontrollable or symptomatic arrhythmias, unstable angina, sick sinus syndrome or second or third degree heart block (unless treated with a permanent, functioning pacemaker), bradycardia (heart rate <55 bpm), and stroke within three months of study screening, and history of myocardial infarction.
* Has Congestive Heart Failure NYHA (New York Heart Association) class II-IV
* Has type 1 diabetes mellitus
* Has newly diagnosed type 2 diabetes (within 4 months of screening visit)
* Has HbA1c > 8.5%
* Has the following, as it relates to subject's antidiabetic therapy:Initiated or changed dosage or formulation of thiazolidinediones (TZDs) within 6 months of screening visit.
* A history of acute or chronic acidosis, including diabetic ketoacidosis
* Has current clinical diagnosis of chronic obstructive pulmonary disease (COPD, e.g., chronic bronchitis) or asthma
* Has a history of bronchospastic disease not undergoing active therapy in whom, in the investigator's opinion, treatment with study medication could provoke bronchospasm
* Has evidence of any of the following clinically significant diseases that could impair the absorption, metabolism, or excretion of orally-administered medication:
* renal disease defined as estimated Glomerular Filtration Rate (eGFR) <60mL/min per 1.73 m2 using the Modification of Diet in Renal Disease (MDRD) formula below: GFR (mL/min/1.73m2) = 186 x [Serum Creatinine (umol/L) x 0.0113]-1.154 x Age(years)-0.203 (x 0.742 if female)
* hepatic disease (i.e., ALT or AST levels greater than three times the upper limit of normal range, history of hepatic impairment, or by clinical assessment)
* Chronic biliary disorders
* Has endocrine disorders (e.g., pheochromocytoma, active and untreated hypo or hyperthyroidism)
* Has any known contraindication to ACE inhibitors, alpha- or beta-blocker treatment
* Has systemic disease, including cancer, with reduced (<12 months) life expectancy
* Has used an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
* Has a history of a psychological illness or any condition that would interfere with the subject's ability to understand or complete the requirements of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, PhD, Principal Investigator — Kaleida Health / University at Buffalo
Locations (1):
- Diabetes - Endocrinology Center of Western New York, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carvedilol: carvedilol Experimental arm
  carvedilol CR (controlled release) added to Lisinopril Doses titrated to maintain optimal blood pressure.
- Lisinopril: lisinopril control arm
  Lisinopril dose titrated to maintain optimal blood pressure.
Period: Overall Study
Arm/Group | Carvedilol | Lisinopril
Started | 7 | 7
Completed | 5 | 6
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Carvedilol: carvedilol
  carvedilol: carvedilol
- Lisinopril: lisinopril
  lisinopril: lisinopril
- Total: Total of all reporting groups
Arm/Group | Carvedilol | Lisinopril | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10) | 59 (11) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 35 (3) | 36 (4) | 35 (3)
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 134 (8) | 137 (7) | 136 (7)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 88 (5) | 89 (5) | 89 (4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Brachial Artery Vascular Reactivity
Description: Percent change from baseline in Brachial artery vascular reactivity at 6 months calculated as: (brachial reactivity at 6 months-brachial reactivity at 0 months)/brachial reactivity at 0 month *100
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Carvedilol | Lisinopril
Number analyzed (Participants) | 5 | 6
percentage of change | 28 (20) | 19 (17)

2. Secondary Outcome: Change in Oxidative Stress in Mononuclear Cells (MNC)
Description: Percent change from baseline in Reactive Oxygen species (ROS) generation in MNC at 6 months calculated as: (ROS at 6 months-ROS at 0 months)/ROS at 0 month *100
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Carvedilol | Lisinopril
Number analyzed (Participants) | 5 | 6
percentage of change | -15 (9) | -10 (11)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Carvedilol | Lisinopril
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes